CLINICAL TRIAL: NCT04682418
Title: Feasibility Study of Pedicle Screw Placement in the Spine With the XVISION SPINE System
Brief Title: Pedicle Screw Placement With XVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augmedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF-VAP-002
Record Dates: First submitted 2019-04-05; First posted 2020-12-23 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-12

CONDITIONS: Spine Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- xvision Spine (Experimental)
  Interventions: Device: xvision Spine sytem

INTERVENTIONS:
Device: xvision Spine sytem — pedicle screw placement will be performed using the XVS navigation system
  Other Names: XVS

SUMMARY:
Open label, prospective, single arm, multi-center study. Pedicle screws placement in sacral/lumbar vertebrae will be performed via open procedural technique, by at least two (2) different surgeons, using the XVISION SPINE system.

Pedicle screw placement accuracy will be assessed by two independent, experienced radiologists, using the Gertzbein score.

Subjects will undergo intraoperative 3D scan prior to screws placement to enable 3D model rendering and XVISION SPINE system registration.

Subjects will undergo intraoperative 3D scan post procedure to enable offline scoring of pedicle screw placement using the Gertzbein score.

Surgeons performing the procedures will be requested to fill in usability questionnaires at the end of the procedure

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 - 80 yrs.
2. Subjects with Spondylosis scheduled to undergo an elective short (6 or less consecutive vertebrae) S1-L1 open spinal fixation surgery using pedicle screws.
3. Subjects requiring a posterior approach surgical procedure.
4. Subjects with normal global spinal alignment (coronal, sagittal view) and/ or patients with degenerative spine disorders.

Exclusion Criteria:

1. Subjects with severe Osteoporosis (T score <-3.5)
2. Subjects with kyphosis at the operated area (≥ stage 3)
3. Subjects with Spondylolisthesis Grade III and above.
4. Subjects scheduled for revision fusion surgery (prior laminectomy or discectomy is not excluded).
5. Subjects with significant abnormalities of bones (e.g. osteogenesis imperfecta, tumors, infection or malignancy, etc.)
6. Subjects with neurologic diseases or damage (e.g. due to trauma, tumor, Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, spina bifida or neurofibroma)
7. Subjects with spinal cord abnormalities with any neurologic symptoms or signs
8. Paraplegia.
9. Pedicle fracture documented before or during surgery.
10. Women pregnant or lactating
11. Subjects requiring anterior release or instrumentation.
12. Subjects who are unwilling to sign written informed consent and assent to participate in the study.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
accurate placement of pedicle screws | through study completion , an average of 6 months.
  accurate placement will be evaluated using Gertzbein and Robbins

SECONDARY OUTCOMES:
usability and ease of use of the system: questionnaire | The surgeon fills a questionnaire after the surgery, within 7 days.
  usability will be evaluated by questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Haemek MC, Afula
  - Sheeba Medical Center, Tel Litwinsky
  - Asaf Harofeh, Tzrifin